CLINICAL TRIAL: NCT01360541
Title: Endoscopic Radiofrequency Ablation for Barrett Oesophagus With Low Grade Dysplasia: a Randomised Controlled Trial vs Endoscopic Surveillance
Brief Title: Radiofrequency Ablation for Barrett Oesophagus With Low Grade Dysplasia
Acronym: RF-DBG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081240
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Barrett Oesophagus; Low Grade Dysplasia
Keywords: Barrett oesophagus; Low grade dysplasia; Radiofrequency ablation
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency ablation (Experimental): Endoscopic radiofrequency ablation of BE
  Interventions: Procedure: Endoscopic radiofrequency ablation
- Surveillance (Active Comparator): Endoscopic surveillance and PPI treatment
  Interventions: Other: Endoscopic surveillance

INTERVENTIONS:
Procedure: Endoscopic radiofrequency ablation — HALO device Use of HALO 360° device for the fist procedure and possible use of HALo 90° device for further treatment sessions Treatment zone of 12cm high maximum. Energy delivered 10 J/cm², power 300W
  Arms: Radiofrequency ablation
Other: Endoscopic surveillance — Upper gastro-intestinal endoscopy every 6 to 12 month under propofol sedation with acetic acid magnification of mucosa and multiple biopsy samples.
  Arms: Surveillance

SUMMARY:
Radiofrequency ablation versus endoscopic surveillance in the management of low grade dysplasia in Barrett oesophagus: a multicentric randomised controlled trial.

DETAILED DESCRIPTION:
Background: The occurrence of low grade dysplasia (LGD) in Barrett oesophagus (BE) is known as a pre-cancerous state. Current recommendation in case of LGD is a close endoscopic surveillance every 6 to 12 month and continuous Proton pomp inhibitor (PPI) treatment. Endoscopic radiofrequency ablation (RFA) has been demonstrated as an efficient treatment to eradicate high grade dysplasia (HGD) and most of LGD and BE.

Main aim of this study: To demonstrate that the prevalence of patients with LGD 3 years after a RFA treatment is lower than in a surveillance group.

Patients & Methods: French multicentric randomized controlled trial for patients with BE with confirmed LGD: RFA vs endoscopic surveillance.

120 patients are planned to be included for at least 40 patients randomized in each group.

Primary endpoint: Prevalence of LGD in each group 3 years after randomization

Secondary endpoints:

* Prevalence of LGD in each group 1 and 5 years after randomization
* Rate of complete eradication of BE at 1, 3 and 5 years after randomization
* Incidence of HGD and adenocarcinoma at 3, 5 years after randomization
* Rate of complications in RFA group after randomization
* Cost - efficacy comparison of the 2 strategies

ELIGIBILITY:
Inclusion Criteria:

* BE with certain LGD in at least one endoscopic biopsy sample
* BE with maximal length of 12cm (Prague classification ≤ C12)
* BE with minimal length of 1cm circumferentially or 3cm in case of a unique zone (Prague classification ≥ C1 or C0M3)
* Patients aged between 18 and 80 years
* Patients' consent for study enrollment
* No contra-indications to general anaesthesia
* Patients ability to take PPI oral medication
* Patient affiliated to a social security system
* No pregnancy and active contraceptions for women in age to procreate
* In case of previous endoscopic mucosal resection for HGD in BE: at least one year of surveillance and 2 biopsy series with LGD without HGD

Exclusion Criteria:

* BE length > 12cm or < 1cm circumferentially (< C1) or < 3cm focally (<M3)
* HGD or adenocarcinoma needing a specific endoscopic or surgical treatment
* Active peptic oesophagitis (Savary III or IV)
* Presence of surgical staples on the area to be treated
* Radiation oesophagitis of radiotherapy whose field includes the lower oesophagus
* previous oesophagus cancer
* previous endoscopic destruction treatment such as photodynamic therapy or plasma argon coagulation
* previous Heller surgery
* oesophagus stenosis
* oesophagus varices
* oesophagus pathology associated with sclerodermia
* Severe coagulation disorders or thrombopenia
* Anaesthesia contra-indications (ASA 4)
* Hypersensitivity to fluorescein or any component of the fluorescein
* Life expectancy < 2 years
* Disability to take PPI oral medication or follow the protocol surveillance Schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of low grade dysplasia 3 years after randomization | 3 years after randomization

SECONDARY OUTCOMES:
Prevalence of low grade dysplasia in each group | 1 and 5 years after randomization
Rate of complete eradication of Barrett oesophagus | 1, 3 and 5 years after randomization
Incidence of high grade dysplasia and adenocarcinoma | 3, 5 years after randomization
Cost - efficacy comparison of the 2 strategies | 5 years
Rate of complications in radiofrequency ablation group | 5 years after randomization
Detection rate of dysplasia and Barrett's oesophagus with the confocal endomicroscopy technique | before treatment, during treatment (Month 3, Month 6, Month 9, Month 12) and after treatment (1, 3 and 5 years after randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic PRAT, MD, PhD, Principal Investigator — Gastroenterology and Endoscopy department, Cochin Hospital
Locations (1):
- Gastroenterology and Endoscopy department, Cochin Hospital, Paris, France

REFERENCES:
- [Background] Barret M, Pioche M, Terris B, Ponchon T, Cholet F, Zerbib F, Chabrun E, Le Rhun M, Coron E, Giovannini M, Caillol F, Laugier R, Jacques J, Legros R, Boustiere C, Rahmi G, Metivier-Cesbron E, Vanbiervliet G, Bauret P, Escourrou J, Branche J, Jilet L, Abdoul H, Kaddour N, Leblanc S, Bensoussan M, Prat F, Chaussade S. Endoscopic radiofrequency ablation or surveillance in patients with Barrett's oesophagus with confirmed low-grade dysplasia: a multicentre randomised trial. Gut. 2021 Jun;70(6):1014-1022. doi: 10.1136/gutjnl-2020-322082. Epub 2021 Mar 8. PMID 33685969